CLINICAL TRIAL: NCT03493880
Title: The Analysis of Immuno-Nutrition Index in Advanced Gastric Cancer Receiving Preoperative Treatments: Observational Cohort Study
Brief Title: The Analysis of Immuno-Nutrition Index in Advanced Gastric Cancer Receiving Preoperative Treatments
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shuang-xi Li, Associate Chief Surgeon, Peking University
Other Study IDs: INdex
Record Dates: First submitted 2018-03-22; First posted 2018-04-11 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Gastric Cancer; Neoadjuvant Chemotherapy; Neoadjuvant Chemoradiotherapy; Systemic Inflammatory Response Syndrome (SIRS); Nutrition Aspect of Cancer
MeSH Terms: conditions — Stomach Neoplasms; Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- naCT: Advanced gastric cancer or esophagogastric cancer receiving neoadjuvant (preoperative) chemotherapy.
- naCRT: Advanced gastric cancer or esophagogastric cancer receiving neoadjuvant (preoperative) chemoradiotherapy.

SUMMARY:
Based on multiple studies, the immune (systemic inflammation) and nutrition index were correlated with short- and long-term prognosis for gastric cancer. With the increasing application of preoperative treatments (chemotherapy and chemoradiotherapy), the issues concerning how are the immuno-nutrition index be altered under the effects of perioperative treatments and what are the clinical values of these index should be clarified.

DETAILED DESCRIPTION:
The immune (systemic inflammation) index includes:

NLR (Neutrophil-to-Lymphocyte Ratio); PLR (Platelet-to-Lymphocyte Ratio); SII (Systemic Immune-Inflammation Index); GPS (Glasgow Prognostic Score); mGPS (modified Glasgow Prognostic Score); PI (Prognostic Index);

The nutrition index includes:

NRS2002; PNI (Prognostic Nutrition Index);

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma
* Received neoadjuvant (preoperative) chemotherapy or chemoradiotherapy
* Diagnosed clinical advanced gastric cancer or esophagogastric cancer

Exclusion Criteria:

* Lack of immuno-nutrition data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the patients with advanced gastric cancer or esophagogastric cancer receiving neoadjuvant chemotherapy or chemoradiotherapy will be included for this observational study.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2015-09-01 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Pathological response | One month after surgery
  Pathological response

SECONDARY OUTCOMES:
3-years overall survival | Three years after surgery
  3-years overall survival
3-years disease-free survival | Three years after surgery
  3-years disease-free survival
Postoperative morbidity | One month after surgery
  Postoperative morbidity
yp TNM Stage | One month after surgery
  yp TNM Stage

CONTACTS AND LOCATIONS:
Overall Officials: Jiafu Ji, M.D., Ph.D., Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China